CLINICAL TRIAL: NCT06596811
Title: Research on the Risk Warning Model and Prevention Strategies for Acute Kidney Injury Associated With Cyclosporine Based on Explainable Deep Neural Networks and Therapeutic Drug Monitoring
Status: Active, not recruiting | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Xiao Li，MD, Associate professor of pharmacy, Qianfoshan Hospital
Other Study IDs: LCYX-LX-20240103
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: AKI; Therapeutic Drug Monitoring (TDM)
Keywords: deep learning; AKI; ADM

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, the investigators will focus on hospitalized patients using cyclosporine and develop an acute kidney injury risk prediction model through in-depth analysis of electronic medical record data, employing interpretable deep learning methods. This model aims to provide timely decision-making support for clinicians regarding prevention and treatment. Compared to traditional machine learning models, deep neural network models can extract deeper features from complex medical data and perform more precise pattern recognition, thereby improving the accuracy and reliability of predictions. By developing a prediction tool based on interpretable deep learning models, the investigators will be able to better assess the association between the use of CNI-class immunosuppressants and acute kidney injury, explore targeted prevention strategies, and offer more accurate prediction and intervention guidance for clinicians. Additionally, this study has significant socioeconomic benefits and promising prospects for application and promotion.

ELIGIBILITY:
Inclusion Criteria:

1. During hospitalization, tacrolimus or cyclosporine was used, and therapeutic drug monitoring was conducted according to standard procedures.
2. Aged 18 years or older at the time of admission.
3. Length of hospital stay > 48 hours.
4. At least 2 serum creatinine tests were conducted during hospitalization.

Exclusion Criteria:

1. Chronic kidney disease stage 5 was achieved before admission.
2. Incomplete clinical data.
3. Serum creatinine levels were consistently below 40 mmol/L during hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inpatients treated with tacrolimus or cyclosporine and monitored for therapeutic drug concentrations at three medical centers from January 2020 to December 2023, including Shandong First Medical University Affiliated Hospital, Binzhou Medical University Affiliated Hospital, and Jinan First People's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
AKI | From January 2020 to December 2023
  Acute kidney injury occurred in hospitalized patients treated with cyclosporine

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Li, Principal Investigator — Qianfoshan Hospital
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, Jinan, China